CLINICAL TRIAL: NCT02715284
Title: A Phase 1 Dose Escalation and Cohort Expansion Study of TSR-042, an Anti-PD-1 Monoclonal Antibody, in Patients With Advanced Solid Tumors
Brief Title: Study of TSR-042, an Anti-programmed Cell Death-1 Receptor (PD-1) Monoclonal Antibody, in Participants With Advanced Solid Tumors
Acronym: GARNET
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 213346; 4010-01-001 (Other: Tesaro)
Record Dates: First submitted 2016-03-09; First posted 2016-03-22 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: Metastatic solid tumors; Advanced solid tumors; Anti-PD-1; TSR-042; Immunotherapy; PD-1; Endometrial; Non-small cell lung cancer; NSCLC; MSI-High; Dostarlimab; dMMR
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Part 1: Participants receiving dostarlimab (Experimental): Part 1 will evaluate dostarlimab at ascending weight-based doses 1 mg/kg, 3 mg/kg and 10 mg/kg. Higher dose levels 15 mg/kg and/or 20 mg/kg may also be explored. Dostarlimab will be administered intravenously (IV) on Day 1 and Day 15 of each cycle; cycle length is 28 days. Cohorts will be enrolled sequentially and will initially follow a 3+3 design.
  Interventions: Biological: Dostarlimab
- Part 2A: Participants receiving dostarlimab (Experimental): In Part 2A, participants will receive fixed dose of 500 mg administered Q3W or 1000 mg administered Q6W dose on Day 1 of each cycle. Cycle duration for Q3W dosing is 21 days and Q6W dosing is 42 days. Cohorts will enroll participants with advanced solid tumor using a modified 6+6 design and will follow a 6+6 design.
  Interventions: Biological: Dostarlimab
- Part 2B: Cohort A1 dMMR/MSI-H endometrial cancer (Experimental): Part 2B: Cohort A1 will include participants with mismatch repair deficient microsatellite instability high (dMMR/MSI-H) endometrial cancer who have progressed on or after platinum doublet therapy. These participants will receive dostarlimab 500 mg for Q3W for the first 4 cycles followed by 1000 mg Q6W for all subsequent cycles. Participants have received no more than 2 lines of anti-cancer therapy for recurrent or advanced (Stage >= IIIB) disease.
  Interventions: Biological: Dostarlimab
- Part 2B: Cohort A2 MMR-proficient/MSS endometrial cancer (Experimental): Part 2B: Cohort A2 will include participants with MMR-proficient/MSS endometrial cancer who have progressed on or after platinum doublet therapy. These participants will receive dostarlimab 500 mg for Q3W for the first 4 cycles followed by 1000 mg Q6W for all subsequent cycles. Participants have received no more than 2 lines of anti-cancer therapy for recurrent or advanced (Stage >=IIIB) disease.
  Interventions: Biological: Dostarlimab
- Part 2B: Cohort E NSCLC (Experimental): Part 2B: Cohort E NSCLC will include participants with non-small cell lung cancer (NSCLC) who progressed after at least 1 prior platinum-based systemic chemotherapy regimen for recurrent or advanced disease. These participants will receive dostarlimab 500 mg for Q3W for the first 4 cycles followed by 1000 mg Q6W for all subsequent cycles.
  Interventions: Biological: Dostarlimab
- Part 2B: Cohort F non-endometrial dMMR/MSI-H or POLE-Mut cancers (Experimental): Participants with recurrent or advanced dMMR/MSI-H solid tumors except endometrial cancers, and gastrointestinal cancers, who have received prior systemic therapy and, who have no alternative treatment options. These participants will receive dostarlimab 500 mg for Q3W for the first 4 cycles followed by 1000 mg Q6W for all subsequent cycles.
  Interventions: Biological: Dostarlimab
- Part 2B: Cohort G PROC without known BRCA (Experimental): Participants with advanced, relapsed, high-grade serous, endometrioid, or clear cell ovarian, fallopian tube, or primary peritoneal cancer without known breast cancer susceptibility gene (BRCA) mutation who have platinum-resistant disease receiving dostarlimab and who have also been previously treated with bevacizumab. These participants will receive dostarlimab 500 mg for Q3W for the first 4 cycles followed by 1000 mg Q6W for all subsequent cycles.
  Interventions: Biological: Dostarlimab

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab (160 mg, 20 mg/mL; or 500 mg, 50 mg/mL) is a humanized monoclonal antibody that binds with high affinity to PD-1 resulting in inhibition of binding to programmed death receptor ligands 1 and 2 (PD-L1 and PD-L2). Dostarlimab will be administered via a 30 minute IV infusion on Day 1 and Day 15 of each cycle in Part 1. For additional patients enrolled specifically to better characterize the PK/PDy profile in Part 1, dostarlimab administration during Cycle 1 will only occur on Day 1 with the second dose administered on Cycle 2/Day 1 and Q2W thereafter. For Part 2A and 2B, dostarlimab will be administered on Day 1 of each treatment cycle. Cycle duration for Q3W dosing is 21 days and Q6W dosing is 42 days.

SUMMARY:
This is a multi-center, open-label, first-in-human Phase 1 study evaluating the anti-programmed death receptor 1 (anti-PD-1) antibody dostarlimab (also known as TSR-042) n participants with advanced solid tumors who have limited available treatment options. The study will be conducted in 2 parts with Part 1 consisting of safety evaluation, pharmacokinetics (PK), and pharmacodynamics (PDy) of escalating doses of dostarlimab. Dose escalation will be based on ascending weight-based dose levels (DLs) of dostarlimab and will continue until the maximum tolerated dose (MTD) is reached or may be stopped at any dose level up to the highest dose of 20 milligrams per kilograms (mg/kg) based on emerging safety and PK/PDy data. Part 2 will be conducted in two subparts, Part 2A (fixed-dose safety evaluation cohorts) and Part 2B (expansion cohorts). Part 2A of the study will evaluate the safety and tolerability of dostarlimab at fixed doses of 500 mg administered every 3 weeks (Q3W) and 1000 mg administered every 6 weeks (Q6W). Part 2B of the study will examine the safety and clinical activity of dostarlimab in cohorts of participants with specific types of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age.
* Participant has proven recurrent or advanced solid tumor and has disease progression after treatment with available anticancer therapies, or is intolerant to treatment that meets the following requirements for the part of the study they will participate in:

A. Part 1: Any histologically or cytologically proven recurrent or advanced solid tumor B. Part 2A: : Any histologically or cytologically proven recurrent or advanced solid tumor

C. Part 2B: Histologically of cytologically proven recurrent or advanced solid tumor with measurable lesion(s) per RECIST version 1.1 and meets one of the following disease types:

The criteria below should be met for participant participating in: 1) Cohort A1 (dMMR/MSI-H endometrial cancer) and 2) Cohort A2 (MMR-proficient/MSS endometrial cancer)

* Participants who have progressed on or after platinum doublet therapy
* Participants have received no more than 2 lines of anticancer therapy for recurrent or advanced (>=Stage IIIB) disease. Prior treatment with hormone therapies is acceptable and does not count towards the number of anticancer therapies noted in the criterion above for this cohort.
* All endometrial cancer histologies are allowed except endometrial sarcoma (including carcinosarcoma).
* Participants must submit 2 scans demonstrating increase in tumor measurement that meet criteria for PD on or after the latest systemic anticancer therapy based on RECIST Version 1.1 to Central Radiology prior to the first dose of dostarlimab.
* Presence of at least 1 measurable lesion on Baseline scan will be confirmed by central radiology review.
* Status of tumor MMR/MSI: Participants can be screened based on local MMR/MSI testing results using immunohistochemistry (IHC), polymerase chain reaction (PCR), or next generation sequencing (NGS) performed in a certified local laboratory, but participant eligibility needs to be determined by MMR IHC results. For participant with available local MMR IHC results for the respective cohort(s), tumor samples have to be submitted to a central IHC laboratory and its quality has to be checked and cleared prior to Cycle 1 Day 1 (C1D1). For participants without available local MMR IHC test results (participants with local PCR or NGS test results), central IHC results have to confirm eligibility prior to proceeding with other screening procedures. After the central IHC test is completed, remaining tumor tissue may be tested for further exploratory biomarkers or may be sent to a central NGS laboratory for further testing.

  3) Cohort E - Participants with NSCLC who progressed after at least 1 prior platinum-based systemic chemotherapy regimen for recurrent or advanced disease.
* Chemotherapy regimen in the adjuvant or neoadjuvant setting following surgery and/or radiation is acceptable if recurrent or advanced disease develops within 6 months from completion of therapy.
* Participants with a known epidermal growth factor receptor (EGFR) mutation must have received a chemotherapy regimen and an EGFR tyrosine kinase inhibitor (TKI) (e.g., erlotinib, gefitinib, afatinib, or experimental)
* Participants with a known anaplastic lymphoma kinase (ALK) translocation must have received a chemotherapy regimen and an ALK inhibitor (e.g., crizotinib, ceritinib or experimental) 4) Cohort F - Participants with recurrent or advanced dMMR/MSI-H solid tumors except endometrial cancers and gastrointestinal cancers, who have received prior systemic therapy and who have no alternative treatment options. Prior treatment with hormone therapies alone given for recurrent or advanced disease is acceptable.
* Presence of at least 1 measurable lesion by RECIST 1.1 on baseline scan will be confirmed by central radiology review prior to first dose of dostarlimab. Patients with primary central nervous system (CNS) tumor should provide brain MRI at baseline.
* Presence of deficient mismatch repair (dMMR) and/or microsatellite instability (MSI-H) in the tumor defined by either:

  i) deficient DNA mismatch repair (dMMR); MMR status must be assessed by immunohistochemistry (IHC) for MMR protein expression (MLH1, MSH2, MSH6, PMS2) where loss of one or more proteins indicates dMMR; dMMR may be determined either locally or by the central reference lab; OR ii) Microsatellite instability (MSI-H); MSI-H as determined by polymerase chain reaction (PCR) or by tissue NGS; MSI-H may be determined locally 5) Cohort G: Participants must have recurrent high-grade serous, endometrioid, or clear cell ovarian, fallopian tube, or primary peritoneal cancer.
* Participants must have presence of at least 1 measurable lesion on Baseline scan that will be confirmed by central radiology review.
* Participants must be considered resistant to the last administered platinum therapy, that is, the time from the last administered platinum dose until the initial documented progression (as evidenced by radiographic progression per RECIST version 1.1) must be less than 6 months.
* Participants must have completed at least 1 but no more than 3 prior lines of therapy for advanced or metastatic ovarian cancer. Neoadjuvant, adjuvant, and the combination of both will be considered as 1 line of therapy. Treatment with single-agent bevacizumab given as maintenance is not counted as a separate line of therapy. If a therapeutic regimen is modified or changed for a reason other than lack of response or PD (such as allergic reaction, toxicity, or drug availability), this is not counted as a separate line of therapy. The use of single-agent hormonal therapy given for reasons other than PD per RECIST version v1.1 (i.e., hormonal therapy given for increasing Cancer antigen [CA]-125 levels) is not counted as a separate line of therapy.
* Participants must have been previously treated with platinum-based regimn, taxane agent(s), and bevacizumab (bevacizumab could be used as a single agent or in combination with another agent, in frontline therapy, as maintenance, or for treatment of recurrent disease).

  • Part 2B: Participants must have archival tumor tissue available that is formalin-fixed and paraffin-embedded (FFPE).
* For participants who do not have archival tissue, a new biopsy must be performed to obtain a tissue sample prior to study treatment initiation. For participants without available archival tissue, the biopsy should be taken from the tumor lesions (either primary or metastatic) that have easy accessibility and low biopsy-associated risks and will exclude biopsies of the liver, brain, lung/mediastinum, pancreas, or endoscopic procedures extending beyond the esophagus, stomach or bowel.
* For Cohort F an FFPE tissue sample must be submitted to the central laboratory for testing. Specimens containing bone are not acceptable. For patients with available local MMR/MSI-H results, tumor samples have to be submitted to a central laboratory and its quality has to be checked and cleared prior to C1D1
* For Cohort G, participant must provide formalin fixed paraffin embedded (FFPE) tumor tissue block(s) with sufficient tumor content (as confirmed by the Sponsor's designated central laboratory) during screening to enable, for example, measures of homologous recombination pathway defects and PD-L1 status. The use of slides created from paraffin-embedded tissue as opposed to FFPE blocks must be approved by the Sponsor.

  • Female participants must have a negative serum pregnancy test within 72 hours prior to the date of the first dose of study medication: unless they are of non-child bearing potential.Non child bearing potential is defined as:
* >= 45 years of age and has not had menses for > 1 year;
* Amenorrheic for < 2 years without a hysterectomy and oophorectomy and have a follicle- stimulating hormone (FSH) value in the postmenopausal range upon pre-study (screening) evaluation.
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound, magnetic resonance imaging (MRI) or computed tomography (CT) scan. Tubal ligation must be confirmed with medical records of the actual procedure.

  * Female participants of childbearing potential must agree to use 1 highly effective form of contraception with their partner starting with the screening visit through 150 days after the last dose of study therapy.
  * Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of <= 2 for Part 1 and <= 1 for Part 2.
  * Participant has an adequate organ function.
  * Participants with known human immunodeficiency virus (HIV) infection are allowed with following requirements:
* Documented evidence of plasma HIV-1 RNA persistently <50 copies (c)/mL ≤3 months prior to AND at Screening. In the >3 to 12 months prior to Screening, plasma HIV-1 RNA consistently <50 c/mL required; if single increases ≥50 c/mL occurred, they cannot have been persistent nor associated with antiretroviral resistance per Investigator's assessment AND
* CD4 cell count >350 cells/mm^3 over past 12 months and at Screening (and no measurement ≤200 cells/mm3 during that time period) AND
* Must be on an uninterrupted combination antiretroviral therapy regimen for at least 3 months prior to Screening, with combination antiretroviral therapy regimen consistent with locally recommended guidelines

  * Participants with history of Centers for Disease Control and Prevention (CDC) Stage 3 disease (CDC, 2014; also known as acquired immunodeficiency syndrome [AIDS]- defining disease) are allowed if AIDS-defining disease has been treated and cured or is stable for ≥3 months prior to study entry. Cutaneous Kaposi's Sarcoma not requiring systemic therapy is allowed.
  * No history of HIV-associated non-Hodgkin lymphoma ≤5 years prior to study and no history of HIV-associated invasive cervical cancer
  * No treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.

Exclusion Criteria:

* Participant has received prior therapy with an anti- programmed death receptor 1 (anti-PD-1), anti-PD-1- ligand-1 (anti-PD-L1), or anti-PD-1 ligand-2 (anti-PD- L2) agent.
* Participant has a known uncontrolled CNS metastasis and/or carcinomatous meningitis.
* Participant has a known additional malignancy that progressed or required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin, squamous cell cancer (SqCC) of the skin that has undergone potentially curative therapy, or in situ cervical cancer, or other neoplastic condition which has undergone curative therapy and is considered cured by the investigator.
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active infection requiring systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled ventricular arrhythmia; recent (within 90 days) myocardial infarction; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent).
* Participant is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the Screening Visit through 150 days after the last dose of study treatment.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Participant has a documented presence of hepatitis B surface antigen [HBsAg] at screening or within 3 months prior to the first dose of study intervention. Participants with a negative HbsAg and positive hepatitis B virus core antibody (HBcAb) result are eligible only if HBV DNA is negative.
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease- modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Use of inhaled steroids, local injection of steroids, and steroid eye drops are allowed.
* Participant has as history of interstitial lung disease.
* Participant has not recovered (i.e., to <= Grade 1 or to Baseline) from radiation- and chemotherapy-induced AEs or received transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte-colony stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 3 weeks prior to the first dose of study drug.
* Participant has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study drug.
* Participant has received prior anticancer therapy (chemotherapy, targeted therapies, radiotherapy, or immunotherapy) within 21 days prior to study Day 1
* Participant has not recovered adequately (<= Grade 1) from AEs and/or complications from any major surgery prior to starting therapy.
* Participant has received a live vaccine within 14 days of planned start of study therapy.
* Participant has a known hypersensitivity to dostarlimab components or excipients.
* For Cohort G, participants will not be eligible if they meet the following criteria:

  * Participants who experienced disease progression within 3 months (as evidenced by radiographic progression per RECIST) of first-line platinum therapy.
  * Participants with known deleterious or suspicious deleterious mutation in BRCA1 or BRCA2 genes (local testing permitted).
  * Participants has received prior therapy with a poly(adenosine diphosphate-ribose) polymerase (PARP)-1/PARP-2 inhibitor.
  * Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, might interfere with the participant's participation for the full duration of the study treatment, or is not in the best interest of the participant to participate.
  * Participant is immunocompromised. Participants with splenectomy are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with treatment emergent AEs (TEAEs) | Up to 2 years
  An adverse event (AE) is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including clinically significant abnormal laboratory findings), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the product. TEAEs defined as any AE either reported for the first time or worsening of a pre-existing event after first dose of study treatment.
Part 1: Number of participants with immune mediated AEs of interest | Up to 2 years
  Participants with immune related AEs of interest will be assessed.
Part 1: Number of participants with abnormal hematology parameters | Up to 2 years
  Blood samples will be collected to assess the following hematology parameters: hemoglobin, Mean corpuscular (MCV), white blood cell count (WBC count), platelets, mean platelet volume, differential WBC count and coagulation factors including International normalized ratio (INR), activated partial thromboplastin time (aPTT) and prothrombin time (PT).
Part 1: Number of participants with abnormal clinical chemistry parameters | Up to 2 years
  Blood samples will be collected to assess the following chemistry parameters: sodium, potassium, calcium, magnesium, creatinine, bilirubin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and albumin.
Part 1, Part 2A, and Part 2B: Number of participants with a change from baseline in urinalysis parameters | Up to 2 years
  Number of participants will be assessed.
Part 1, Part 2A, and Part 2B: Number of participants with a change from baseline in vital signs | Up to 2 years
  Number of participants will be assessed.
Part 1: Number of participants with abnormal electrocardiogram (ECG) parameters | Up to 2 years
  Participants will be supine or in a semi-recumbent position and rested for approximately 2 minutes before ECGs are recorded.
Part 1: Number of participants receiving concomitant medications | Up to 2 years
  Concomitant medications will be recorded.
Part 2A: Number of participants with TEAEs | Up to 2 years
  An AE is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including clinically significant abnormal laboratory findings), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the product. TEAEs defined as any AE either reported for the first dose of study treatment.
Part 2A: Number of participants with immune mediated AEs of interest | Up to 2 years
  Participants with immune related AEs of interest will be assessed.
Part 2A: Number of participants with abnormal hematology parameters | Up to 2 years
  Blood samples will be collected to assess the following hematology parameters: hemoglobin, MCV, white WBC count, platelets, mean platelet volume, differential WBC count and coagulation factors including INR, aPTT and PT.
Part 2A: Number of participants with abnormal clinical chemistry parameters | Up to 2 years
  Blood samples will be collected to assess the following chemistry parameters: sodium, potassium, calcium, magnesium, creatinine, bilirubin, AST, ALT, and albumin.
Part 2A: Number of participants with abnormal ECG | Up to 2 years
  Participants will be supine or in a semi-recumbent position and rested for approximately 2 minutes before ECGs are recorded.
Part 2A: Number of participants receiving concomitant medications | Up to 2 years
  Concomitant medications will be recorded.
Part 2B: Number of participants with TEAEs | Up to 2 years
  An AE is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including clinically significant abnormal laboratory findings), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the product. TEAEs defined as any AE either reported for the first dose of study treatment.
Part 2B: Number of participants with immune related AEs of interest | Up to 2 years
  Participants with immune related AEs of interest will be assessed.
Part 2B: Number of participants with abnormal hematology parameters | Up to 2 years
  Blood samples will be collected to assess the following hematology parameters: hemoglobin, MCV, white WBC count, platelets, mean platelet volume, differential WBC count and coagulation factors including INR, aPTT and PT.
Part 2B: Number of participants with abnormal clinical chemistry parameters | Up to 2 years
  Blood samples will be collected to assess the following chemistry parameters: sodium, potassium, calcium, magnesium, creatinine, bilirubin, AST, ALT, and albumin.
Part 2B: Number of participants with abnormal ECG parameters | Up to 2 years
  Participants will be supine or in a semi-recumbent position and rested for approximately 2 minutes before ECGs are recorded.
Part 2B: Number of participants receiving concomitant medications | Up to 2 years
  Concomitant medications will be recorded.
Part 2B: Cohort A1 Overall Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 2 years
  ORR is defined as the proportion of participants achieving complete response (CR) or partial response (PR) as evaluated by independent blinded central review using RECIST version 1.1.
Part 2B: Cohort F ORR by RECIST version 1.1 | Up to 2 years
  ORR is defined as the proportion of participants achieving CR or PR as evaluated by independent blinded central review using RECIST version 1.1.
Part 2B: Cohort A2 ORR by RECIST version 1.1 | Up to 2 years
  ORR is defined as the proportion of participants achieving CR or PR as evaluated by independent blinded central review using RECIST version 1.1.
Part 2B: Cohort G ORR by RECIST version 1.1 | Up to 2 years
  ORR is defined as the proportion of participants achieving CR or PR as evaluated by independent blinded central review using RECIST version 1.1.
Part 2B: Cohort E ORR by immune related Response Evaluation Criteria in Solid Tumors per irRECIST | Up to 2 years
  ORR is defined as the proportion of participants achieving CR or PR as assessed by investigator per irRECIST will be evaluated.
Part 2B: Cohort A1 Duration of response (DOR) | Up to 2 years
  DOR is defined as the time from first documentation of CR or PR by RECIST version 1.1 until the time of first documentation of progressive disease (PD) evaluated using RECIST version 1.1 based on independent blinded central review, or death due to any cause.
Part 2B: Cohort F Duration of response (DOR) | Up to 2 years
  DOR is defined as the time from first documentation of CR or PR by RECIST version 1.1 until the time of first documentation of PD evaluated using RECIST version 1.1 based on independent blinded central review, or death due to any cause.
Part 2B: Cohort A2 Duration of response (DOR) | Up to 2 years
  DOR is defined as the time from first documentation of CR or PR by RECIST version 1.1 until the time of first documentation of PD evaluated using RECIST version 1.1 based on independent blinded central review, or death due to any cause.

SECONDARY OUTCOMES:
Part 1: Immune-related objective response rate (irORR) by irRECIST | Up to 2 years
  Immune-related objective response rate will be evaluated based on investigator's assessment using irRECIST.
Part 2B: Cohort A1 ORR by independent blinded central review using RECIST version 1.1 | Up to 2 years
  ORR is defined as the proportion of participants achieving CR or PR as evaluated by independent blinded central review using RECIST version 1.1.
Part 2B: Cohort F ORR by independent blinded central review using RECIST version 1.1 | Up to 2 years
  ORR is defined as the proportion of participants achieving CR or PR as evaluated by independent blinded central review using RECIST version 1.1.
Part 2B: Cohort A1 Immune-related objective response rate (irORR) by irRECIST | Up to 2 years
  Immune related objective response rate will be evaluated based on investigator's assessment using irRECIST.
Part 2B: Cohort A2 irORR by irRECIST | Up to 2 years
  Immune related objective response rate will be evaluated based on investigator's assessment using irRECIST.
Part 2B: Cohort F irORR by irRECIST | Up to 2 years
  Immune related objective response rate will be evaluated based on investigator's assessment using irRECIST.
Part 2B: Cohort G irORR by irRECIST | Up to 2 years
  Immune related objective response rate will be evaluated based on investigator's assessment using irRECIST.
Part 2B: Cohort A1 Duration of response (DOR) based on independent blinded central review using RECIST version 1.1 | Up to 2 years
  DOR is defined as the time from first documentation of CR or PR by RECIST version 1.1 until the time of first documentation of progressive disease (PD) evaluated using RECIST version 1.1 based on independent blinded central review, or death due to any cause.
Part 2B: Cohort F DOR based on independent blinded central review using RECIST version 1.1 | Up to 2 years
  DOR is defined as the time from first documentation of CR or PR by RECIST version 1.1 until the time of first documentation of PD evaluated using RECIST version 1.1 based on independent blinded central review, or death due to any cause.
Part 2B: Cohort G DOR based on independent blinded central review using RECIST version 1.1 | Up to 2 years
  DOR is defined as the time from first documentation of CR or PR by RECIST version 1.1 until the time of first documentation of PD evaluated using RECIST version 1.1 based on independent blinded central review, or death due to any cause.
Part 2B: Cohort A1 Disease control rate | Up to 2 years
  Disease control rate is the proportion of participants achieving CR, PR, or SD per RECIST v1.1 based on independent blinded central review.
Part 2B: Cohort A2 Disease control rate | Up to 2 years
  Disease control rate is the proportion of participants achieving CR, PR, or SD per RECIST v1.1 based on independent blinded central review.
Part 2B: Cohort F Disease control rate | Up to 2 years
  Disease control rate is the proportion of participants achieving CR, PR, or SD per RECIST v1.1 based on independent blinded central review.
Part 2B: Cohort G Disease control rate | Up to 2 years
  Disease control rate is the proportion of participants achieving CR, PR, or SD per RECIST v1.1 based on independent blinded central review.
Immune related disease control rate | Up to 2 years
  The proportion of participants achieving CR, PR, or SD per irRECIST based on Investigators assessment.
Immune related duration of response | Up to 2 years
  The time from first documentation of CR or PR by irRECIST until the time of first documentation of PD (subsequently confirmed) per irRECIST based on Investigators assessment.
Progression free survival | Up to 2 years
  The time from date of first dose to the earlier date of assessment of progression or death by any cause in the absence of progression based on: (1) the time of first documentation of PD per RECIST v1.1 (for Cohorts A1, A2, F, and G only); and (2) the time of first documentation of PD (subsequently confirmed) per irRECIST.
Overall survival | Up to 2 years
  The time from date of first dose of study treatment to the date of death by any cause.
Part 1: Area under the concentration-time curve from time 0 to last (AUC,0-last) assessment of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504 and 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Area under the concentration-time curve from time 0 to infinity (AUC, 0-infinity) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Minimum concentration (Cmin) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Maximum concentration (Cmax) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Clearance (CL) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Volume of distribution (Vz) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Area under the concentration-time curve at steady state (AUC,ss) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Minimum concentration at steady state (Cmin,ss) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504,672 hours post dose.
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1: Maximum concentration at steady state (Cmax,ss) of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: AUC,0-last assessment of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504 hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: AUC, 0-infinity of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504 hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Cmin of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504,hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected
Part 2A: Cmax of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504,hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: CL of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504,hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Vz of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504 hours post dose Q3W upto 2 years.
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: AUC,ss of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504 hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Cmin,ss of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504 hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Cmax,ss of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, and 504 hours post dose Q3W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A : AUC,0-last assessment of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: AUC, 0-infinity of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Cmin of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Cmax of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: CL of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Vz of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: AUC,ss of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Cmin,ss of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840, and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2A: Cmax,ss of dostarlimab | Predose, 0.25, 0.5, 1.5, 3, 24, 48, 96, 168, 336, 504, 672, 840 and 1008 hours post dose Q6W upto 2 years
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2B: Cmax of dostarlimab | Predose, 0.5 and 1.5 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2B: AUC,ss of dostarlimab | Predose, 0.5 and 1.5 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 2B: Cmax,ss of dostarlimab | Predose, 0.5 and 1.5 hours post dose
  Blood samples for determination of serum levels of dostarlimab will be collected.
Part 1, Part 2A, and Part 2B: Number of participants with antidrug antibodies (ADA) against dostarlimab | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (41):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Marcos, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Fairway, Kansas
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Farmington, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Jamaica, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Hilliard, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, São Paulo, Brazil
- Canada (8):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Czechia (2):
  - GSK Investigational Site, Hořovice
  - GSK Investigational Site, Zlín
- Denmark (2):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Odense C
- France (6):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Villejuif
- Italy (5):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Naples
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Verona
- Poland (4):
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Torun
- Spain (9):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- United Kingdom (6):
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Patnaik A, Weiss GJ, Rasco DW, Blaydorn L, Mirabella A, Beeram M, Guo W, Lu S, Danaee H, McEachern K, Im E, Sachdev JC. Safety, antitumor activity, and pharmacokinetics of dostarlimab, an anti-PD-1, in patients with advanced solid tumors: a dose-escalation phase 1 trial. Cancer Chemother Pharmacol. 2022 Jan;89(1):93-103. doi: 10.1007/s00280-021-04358-3. Epub 2021 Nov 8. PMID 34750637
- [Background] Zhang XT, Chen H, Shao W, Zhongping JL, Melham M, Lu S.A Competitive Ligand Binding Assay to Measure Antidrug Antibodies Against Dostarlimab (TSR-042).2021; DOI: 10.1186/s41120-021-00039-w
- [Background] Patterson M, Beausang LA, Rup B, Bowsher R, Krug K, Gunn G, Melham M, Lu S.A Bridging Assay for Detection and Characterization of Anti-Drug Antibodies to Dostarlimab, a New Anti-PD-1 Therapeutic Monoclonal Antibody .2021;7(11) DOI: DOI 10.1186/s41120-021-00045-y
- [Background] Kumar S, Ghosh S, Sharma G, Wang Z, Kehry MR, Marino MH, Neben TY, Lu S, Luo S, Roberts S, Ramaswamy S, Danaee H, Jenkins D. Preclinical characterization of dostarlimab, a therapeutic anti-PD-1 antibody with potent activity to enhance immune function in in vitro cellular assays and in vivo animal models. MAbs. 2021 Jan-Dec;13(1):1954136. doi: 10.1080/19420862.2021.1954136. PMID 34313545
- [Background] Oaknin A, Gilbert L, Tinker AV, Brown J, Mathews C, Press J, Sabatier R, O'Malley DM, Samouelian V, Boni V, Duska L, Ghamande S, Ghatage P, Kristeleit R, Leath C III, Guo W, Im E, Zildjian S, Han X, Duan T, Veneris J, Pothuri B. Safety and antitumor activity of dostarlimab in patients with advanced or recurrent DNA mismatch repair deficient/microsatellite instability-high (dMMR/MSI-H) or proficient/stable (MMRp/MSS) endometrial cancer: interim results from GARNET-a phase I, single-arm study. J Immunother Cancer. 2022 Jan;10(1):e003777. doi: 10.1136/jitc-2021-003777. PMID 35064011
- [Background] Kristeleit R, Mathews C, Redondo A, Boklage S, Hanlon J, Im E, Brown J. Patient-reported outcomes in the GARNET trial in patients with advanced or recurrent mismatch repair-deficient/microsatellite instability-high endometrial cancer treated with dostarlimab. Int J Gynecol Cancer. 2022 Oct 3;32(10):1250-1257. doi: 10.1136/ijgc-2022-003492. PMID 35973737
- [Background] Kuchimanchi M, Dabrowski C, Lu S, Melhem M. Dostarlimab, an anti-programmed death-1 monoclonal antibody, does not cause QT prolongation in patients with solid tumours: A concentration-QT analysis. Br J Clin Pharmacol. 2023 Jul;89(7):2272-2282. doi: 10.1111/bcp.15700. Epub 2023 Mar 20. PMID 36823349
- [Derived] Andre T, Berton D, Curigliano G, Sabatier R, Tinker AV, Oaknin A, Ellard S, de Braud F, Arkenau HT, Trigo J, Gravina A, Kristeleit R, Moreno V, Abdeddaim C, Vano YA, Samouelian V, Miller R, Boni V, Torres AA, Gilbert L, Brown J, Dewal N, Dabrowski C, Antony G, Zografos E, Veneris J, Banerjee S. Antitumor Activity and Safety of Dostarlimab Monotherapy in Patients With Mismatch Repair Deficient Solid Tumors: A Nonrandomized Controlled Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2341165. doi: 10.1001/jamanetworkopen.2023.41165. PMID 37917058
- [Derived] Rodrigues M, Eberst L, Follana P, Gauthier L, Jacquemin V, Tessier C, El Mouaddin N, Boudier P, Fiteni F, Angeli E, Roche S, Delanoy N, Sabatier R, Flippot R, de la Motte Rouge T. Real-world dostarlimab use in advanced/recurrent endometrial cancer in France. Bull Cancer. 2023 Oct;110(10):1041-1050. doi: 10.1016/j.bulcan.2023.06.009. Epub 2023 Aug 31. PMID 37659907
- [Derived] Oaknin A, Pothuri B, Gilbert L, Sabatier R, Brown J, Ghamande S, Mathews C, O'Malley DM, Kristeleit R, Boni V, Gravina A, Banerjee S, Miller R, Pikiel J, Mirza MR, Dewal N, Antony G, Dong Y, Zografos E, Veneris J, Tinker AV. Safety, Efficacy, and Biomarker Analyses of Dostarlimab in Patients with Endometrial Cancer: Interim Results of the Phase I GARNET Study. Clin Cancer Res. 2023 Nov 14;29(22):4564-4574. doi: 10.1158/1078-0432.CCR-22-3915. PMID 37363992
- [Derived] Moreno V, Roda D, Pikiel J, Trigo J, Bosch-Barrera J, Drew Y, Kristeleit R, Hiret S, Bajor DL, Cruz P, Beck JT, Ghosh S, Dabrowski C, Antony G, Duan T, Veneris J, Zografos E, Subramanian J. Safety and Efficacy of Dostarlimab in Patients With Recurrent/Advanced Non-small Cell Lung Cancer: Results from Cohort E of the Phase I GARNET Trial. Clin Lung Cancer. 2022 Nov;23(7):e415-e427. doi: 10.1016/j.cllc.2022.05.013. Epub 2022 May 23. PMID 35729005
- [Derived] Oaknin A, Tinker AV, Gilbert L, Samouelian V, Mathews C, Brown J, Barretina-Ginesta MP, Moreno V, Gravina A, Abdeddaim C, Banerjee S, Guo W, Danaee H, Im E, Sabatier R. Clinical activity and safety of the anti-PD-1 monoclonal antibody dostarlimab for patients with recurrent or advanced dMMR endometrial cancer. Future Oncol. 2021 Oct 1;17(29):3781-3785. doi: 10.2217/fon-2021-0598. Epub 2021 Aug 24. PMID 34427115
- [Derived] Oaknin A, Tinker AV, Gilbert L, Samouelian V, Mathews C, Brown J, Barretina-Ginesta MP, Moreno V, Gravina A, Abdeddaim C, Banerjee S, Guo W, Danaee H, Im E, Sabatier R. Clinical Activity and Safety of the Anti-Programmed Death 1 Monoclonal Antibody Dostarlimab for Patients With Recurrent or Advanced Mismatch Repair-Deficient Endometrial Cancer: A Nonrandomized Phase 1 Clinical Trial. JAMA Oncol. 2020 Nov 1;6(11):1766-1772. doi: 10.1001/jamaoncol.2020.4515. PMID 33001143